CLINICAL TRIAL: NCT07172828
Title: Investigation of the Effects of Virtual Reality-Based Rehabilitation on Muscle Architecture, Balance Control, and Patient Satisfaction in Individuals With Chronic Low Back Pain
Brief Title: Virtual Reality-Based Rehabilitation in Chronic Low Back Pain: Effects on Muscle Architecture, Balance, and Satisfaction (VR-LBPREHAB)
Acronym: VR-LBPREHAB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, ABDURAHİM ASLIYÜCE, Principal Investigator, Physiotherapist (MSc), Research Assistant, PhD Candidate, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FTREK25/40
Record Dates: First submitted 2025-08-26; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Chronic Low Back Pain (CLBP); Musculoskeletal Pain; Postural Balance; Exercise Therapy
Keywords: Low Back Pain; Virtual Reality Rehabilitation; Muscle Architecture; Thoracolumbar Fascia; Balance Control; Exercise Therapy
MeSH Terms: conditions — Musculoskeletal Pain; Low Back Pain

STUDY DESIGN:
Intervention Model Description: This study is designed as a two-arm randomized controlled trial with parallel assignment. A total of 40-50 participants with chronic low back pain will be randomly allocated to one of two groups: (1) the experimental group, receiving an 8-week virtual reality (VR)-based rehabilitation program, or (2) the control group, receiving conventional motor control exercises. Each program will be delivered three times per week, 40 minutes per session, for a total of 24 sessions. The parallel assignment model ensures that each participant receives only one type of intervention throughout the study period, allowing for a direct comparison between VR-based rehabilitation and conventional exercise therapy.
Who Masked: Outcomes Assessor
Masking Description: Participants will be randomized into two groups using a sealed-envelope method: a virtual reality group and a conventional rehabilitation group. The VR group will perform 20 minutes of motor control exercises plus 20 minutes of Pilates-based VR games (5 reps/set), while the control group will complete 40 minutes of progressive motor control/stabilization exercises (10 reps/set). Both groups will train 3 times per week for 8 weeks. Ultrasound imaging assessments will be performed by an experienced physiotherapist who will remain blinded to group allocation. This ensures that outcome assessment of muscle architecture is conducted under blinded conditions. Participants and care providers will not be blinded due to the visible nature of the interventions. Evaluations at baseline, 8 weeks, 3 and 6 months will include ultrasound, balance, pain, disability, and patient satisfaction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality-Based Rehabilitation Group (Experimental): Participants receive 20 minutes of motor control exercises combined with 20 minutes of Pilates-based virtual reality games (5 repetitions per set), delivered three times per week for 8 weeks (24 sessions in total).
  Interventions: Behavioral: Virtual Reality-Based Rehabilitation
- Conventional Rehabilitation Group (Active Comparator): Participants perform 40 minutes of progressive spinal stabilization and motor control exercises (10 repetitions per set), delivered three times per week for 8 weeks (24 sessions in total).
  Interventions: Behavioral: Conventional Motor Control Exercises

INTERVENTIONS:
Behavioral: Virtual Reality-Based Rehabilitation — Participants receive 20 minutes of motor control exercises combined with 20 minutes of Pilates-inspired virtual reality games (5 repetitions per set). Training will be delivered three times per week, 40 minutes per session, for 8 weeks (24 sessions in total).
  Other Names: VR-Based Exercise; VR Rehabilitation
  Arms: Virtual Reality-Based Rehabilitation Group
Behavioral: Conventional Motor Control Exercises — Participants perform 40 minutes of progressive spinal stabilization and motor control exercises (10 repetitions per set), three times per week for 8 weeks (24 sessions in total).
  Other Names: Progressive Stabilization Exercises; Standard Exercise Therapy
  Arms: Conventional Rehabilitation Group

SUMMARY:
Chronic low back pain is a common musculoskeletal disorder that causes pain, disability, and reduced quality of life. It is often related to changes in trunk muscle function, thoracolumbar fascia morphology, and impaired balance control. Although conventional motor control exercises are effective, patient motivation and adherence can be limited. Virtual reality (VR)-based rehabilitation offers interactive and engaging environments that may improve compliance and provide additional therapeutic benefits.

This study is a randomized controlled trial designed to investigate the effects of VR-based rehabilitation compared with conventional motor control exercises in individuals with chronic low back pain. A total of 40-50 participants aged 18-65 will be recruited and randomly assigned to one of two groups: (1) VR-based rehabilitation or (2) conventional exercise therapy. Both programs will last 8 weeks, delivered three times per week for 40 minutes per session.

The primary outcomes include muscle architecture assessed by ultrasound imaging, thoracolumbar fascia morphology, and postural balance control measured by force platform tests. Secondary outcomes include pain intensity, disability, fear-avoidance beliefs, quality of life, and patient satisfaction.

The findings of this study are expected to provide new insights into the role of VR in rehabilitation and contribute to evidence-based strategies for managing chronic low back pain. By exploring the effects on both physical and patient-reported outcomes, the study may highlight innovative approaches to improve adherence, reduce pain, and enhance daily function in affected individuals.

DETAILED DESCRIPTION:
Chronic low back pain is a prevalent musculoskeletal condition associated with altered muscle activation, impaired postural control, and thoracolumbar fascia changes that may contribute to persistent pain and disability. Conventional rehabilitation approaches such as stabilization and motor control exercises are widely recommended, yet patient adherence and motivation often limit their effectiveness.

Virtual reality (VR)-based rehabilitation integrates visual, auditory, and interactive elements that can enhance engagement, provide distraction from pain, and encourage more consistent exercise participation. While VR interventions have shown benefits in populations such as stroke, cerebral palsy, and multiple sclerosis, the evidence in chronic low back pain remains limited.

This randomized controlled trial is designed to investigate the clinical and functional effects of VR-based rehabilitation compared with conventional motor control exercises in individuals with chronic low back pain. The intervention will combine traditional physiotherapy approaches with VR-based exercises to evaluate potential improvements in muscle architecture, balance control, and patient-centered outcomes such as satisfaction and adherence.

The study will contribute novel data on the feasibility and effectiveness of VR-based rehabilitation in chronic low back pain, with the goal of providing physiotherapists and clinicians with evidence to guide innovative treatment strategies. The adapted approach is expected to promote adherence, improve functional outcomes, and address gaps in the current literature on VR applications in musculoskeletal rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Chronic low back pain persisting for ≥ 3 months.
* Literacy and Montreal Cognitive Assessment (MoCA) score > 21.
* Voluntary participation with signed informed consent.

Exclusion Criteria:

* Malignancy.
* Pregnancy.
* History of epilepsy (including photosensitive seizures), dementia, migraine, or other neurological disorders limiting VR use.
* Surgery within the past 6 months.
* Received physiotherapy or rehabilitation services in the past 6 months.
* Presence of acute infection.
* Unhealed fracture.
* Withdrawal of informed consent at any stage of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-13 (Estimated); Primary Completion 2026-10-13 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Change in Transversus Abdominis Thickness (mm) | Baseline, 8 weeks, 3 months, 6 months.
  Measured by ultrasound in supine hook-lying position.
Change in Internal Oblique Thickness (mm) | Baseline, 8 weeks, 3 months, 6 months.
  Measured by ultrasound in supine hook-lying position
Change in External Oblique Thickness (mm) | Baseline, 8 weeks, 3 months, 6 months.
  Measured by ultrasound in supine hook-lying position
Change in Rectus Abdominis Thickness (mm) | Baseline, 8 weeks, 3 months, 6 months.
  Measured by ultrasound in supine hook-lying position
Change in Thoracolumbar Fascia Thickness (mm) | Baseline, 8 weeks, 3 months, 6 months.
  Measured bilaterally at L3 level in prone position.
Change in Thoracolumbar Fascia Morphology (categorical) | Baseline, 8 weeks, 3 months, 6 months.
  ssessed bilaterally at L3 level in prone position (regular vs. irregular morphology).
Change in Postural Sway (mm) | Baseline, 8 weeks, 3 months, 6 months.
  Anterior-posterior and medio-lateral sway measured by force platform (Freemed, Sensor Medica).
Change in Limits of Stability (mm/°/s) | Baseline, 8 weeks, 3 months, 6 months.
  Maximum excursion, reaction time, movement velocity, and directional control measured by force platform (Freemed, Sensor Medica).

SECONDARY OUTCOMES:
Pain Intensity | Baseline, 8 weeks, 3 months, 6 months.
  Pain severity measured using the Numeric Pain Rating Scale (0-10).
Functional Disability | Baseline, 8 weeks, 3 months, 6 months.
  Functional status assessed with the Oswestry Disability Index
Functional Disability | Baseline, 8 weeks, 3 months, 6 months.
  Functional status assessed with the Back Performance Scale.
Lumbar Paravertebral Muscle Stiffness (N/m) | Baseline, 8 weeks, 3 months, 6 months.
  Assessed with MyotonPRO at bilateral L5.
Lumbar Paravertebral Muscle Elasticity (ratio) | Baseline, 8 weeks, 3 months, 6 months.
  Assessed with MyotonPRO at bilateral L5.
Trunk Muscle Endurance (mmHg, seconds) | Baseline, 8 weeks, 3 months, 6 months.
  Endurance of the Transversus Abdominis muscle assessed with the Stabilizer Pressure Biofeedback device.
Fear-Avoidance Beliefs | Baseline, 8 weeks, 3 months, 6 months.
  Psychological aspects evaluated using the Fear-Avoidance Beliefs Questionnaire (FABQ).
Change in Quality of Life (Nottingham Health Profile Total Score) | Baseline, 8 weeks, 3 months, 6 months.
  Quality of life assessed using the Nottingham Health Profile (NHP); includes domains of pain, emotional reaction, sleep, social isolation, physical activity, and energy. Higher scores indicate poorer quality of life.
Patient Satisfaction | 8 weeks, 3 months, 6 months.
  Satisfaction levels assessed using the Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST 2.0).
Exercise Adherence | During the 8-week intervention.
  Recorded via exercise diary including weekly frequency and duration of sessions.
Body Composition | Baseline, 8 weeks, 3 months, 6 months.
  Body weight, BMI, and body fat percentage measured using a bioimpedance analyzer (Tanita MC180MA).

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ülger, PT, PhD, Study Director — Hacettepe University, Faculty of Physical Therapy and Rehabilitation; Abdurahim Aslıyüce, Research Assistant, MSc, PT, Principal Investigator — Hacettepe University, Faculty of Physical Therapy and Rehabilitation
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because of privacy and confidentiality considerations. All data will remain anonymized and securely stored, with access restricted to the research team in accordance with ethics committee approval.

REFERENCES:
- [Background] Taguchi T, Tesarz J, Mense S. The thoracolumbar fascia as a source of low back pain. In: Fascia Research II - Basic Science and Implications for Conventional and Complementary Healthcare. Munich: Elsevier GmbH; 2009:251.
- [Background] Li R, Li Y, Kong Y, Li H, Hu D, Fu C, Wei Q. Virtual Reality-Based Training in Chronic Low Back Pain: Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Med Internet Res. 2024 Feb 26;26:e45406. doi: 10.2196/45406. PMID 38407948
- [Background] Brea-Gomez B, Torres-Sanchez I, Ortiz-Rubio A, Calvache-Mateo A, Cabrera-Martos I, Lopez-Lopez L, Valenza MC. Virtual Reality in the Treatment of Adults with Chronic Low Back Pain: A Systematic Review and Meta-Analysis of Randomized Clinical Trials. Int J Environ Res Public Health. 2021 Nov 11;18(22):11806. doi: 10.3390/ijerph182211806. PMID 34831562
- [Background] Hartvigsen J, Hancock MJ, Kongsted A, Louw Q, Ferreira ML, Genevay S, Hoy D, Karppinen J, Pransky G, Sieper J, Smeets RJ, Underwood M; Lancet Low Back Pain Series Working Group. What low back pain is and why we need to pay attention. Lancet. 2018 Jun 9;391(10137):2356-2367. doi: 10.1016/S0140-6736(18)30480-X. Epub 2018 Mar 21. PMID 29573870
- [Background] Hoy D, Bain C, Williams G, March L, Brooks P, Blyth F, Woolf A, Vos T, Buchbinder R. A systematic review of the global prevalence of low back pain. Arthritis Rheum. 2012 Jun;64(6):2028-37. doi: 10.1002/art.34347. Epub 2012 Jan 9. PMID 22231424